CLINICAL TRIAL: NCT04261231
Title: Correlation of the "Preliminary Universal Surgical Invasiveness Score" (pUSIS) With Short Term Post-operative Clinical Outcome Parameters. An Observational Study
Acronym: pUSISoutcome
Status: Completed | Type: Observational
Sponsor: University of Zurich (Other)
Responsible Party: Sponsor
Other Study IDs: BASEC 2016-00498
Record Dates: First submitted 2020-02-06; First posted 2020-02-07 (Actual); Last update posted 2020-04-02 (Actual); Status verified 2020-03

CONDITIONS: Outcome Assessment, Health Care
MeSH Terms: interventions — Surgical Procedures, Operative; Anesthesia

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: Surgery and anesthesia — Elective surgery in adults

SUMMARY:
The scope of this investigation is to demonstrate that the pUSIS values correlate closely with short term post-operative clinical outcome parameters, thus making this scoring system a good predictor for the patients' postoperative course and may become a helpful instrument for decision making concerning the choice of postoperative surveillance and treatment. The obtained follow up results were subjected to correlation analyzis with the pUSIS values in order to determine their association and if possible to recognize threshold values that may indicate a suitable type/intensity of postoperative surveillance.

DETAILED DESCRIPTION:
a number of 60 day-care as well as 100 in-hospital patients undergoing elective surgery in general anesthesia have been enrolled into this observational study. The recruitment of cases happened randomly on a daily basis according to the available operations in the surgical unit where the main investigator (NN) was performing her/his anesthesiological services. Thus there was no selection of specific surgeries or surgical disciplines.

Inclusion criteria: adult patients (>18 y) undergoing surgery in general anesthesia.

Exclusion criteria: emergency cases, patients aged < 18 years, pregnant women, inability to give informed consent.

The data acquisition consisted of calculation of the individual pUSIS for the selected cases by end of surgery, and by collecting in the follow up period the following set of short term parameters:

In-hospital patients

* time duration from end of surgery till discharge from PACU
* time duration from end of surgery till discharge from IMCU
* time duration from end of surgery till discharge from ICU
* time duration from end of surgery till discharge from hospital up to 30 days
* Occurrence and severity of complications the during hospital stay or up to 30 days according to a predefined list

Day-care patients

* time duration from end of surgery till discharge from PACU
* time duration from end of surgery till discharge from hospital
* Occurrence and severity of complications the during hospital stay according to a predefined list
* Occurrence of readmission due to complications within a period of 10 days after surgery

The predefined list of complications that could be observed during the follow up period consists of:

* Occurrence of postoperative pain that needed medical intervention, duration of this state, average severity level (according an ordinal scale with the levels: mild, moderate, severe)
* Occurrence of hemodynamic instability, duration of this state, average severity level (according an ordinal scale with the levels: mild, moderate, severe)
* Occurrence of postoperative hemorrhage, quantification in total ml of estimated blood loss
* Occurrence of respiratory support, duration of this state
* Occurrence of thrombo-embolic complications
* Occurrence of hepato-renal complications
* Occurrence of cerebral/neurological complications
* Occurrence of infectiological/inflamatory complications
* Average level of self-assessed subjective wellbeing (according an ordinal scale with the levels: excellent, rather good, moderate, bad, extremely bad)

The obtained follow up results were subjected to correlation analyzis with the pUSIS values in order to determine their association and if possible to recognize threshold values that may indicate a suitable type/intensity of postoperative surveillance.

ELIGIBILITY:
Inclusion Criteria:

* adult patients (>18 y) undergoing surgery in general anesthesia

Exclusion Criteria:

* emergency cases
* patients aged < 18 years
* pregnant women
* inability to give informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: General surgical patients.
Sampling Method: Non-Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2019-11-01 (Actual); Primary Completion 2020-03-31 (Actual); Study Completion 2020-03-31 (Actual)

PRIMARY OUTCOMES:
Duration of postoperative hospital stay | 1-60 days
  In-hospital days
Duration if intensive care treatment | 600 hours
  ICU hours
Duration of postoperative ventilation | 600 hours
  Ventilation hours
Postoperative complications | 1-60 days
  thromboembolic, hepato-renal, neorologal, infections

SECONDARY OUTCOMES:
Subjective wellbeeing | 1-60 days
  Likert scale 1 (excellent) to 5 (exteremely bad)

CONTACTS AND LOCATIONS:
Locations (1):
- University Hospital Zurich, Institue of Anesthesiology, Zurich, Canton of Zurich, Switzerland

IPD SHARING:
Plan to Share IPD: No
No plan to share.

REFERENCES:
- [Background] Biro P, Gurman G. Proposal for a surrogate surgical invasiveness score to obtain a 'post hoc' quantification of surgical stress and tissue trauma in the context of postoperative outcome assessments. Br J Anaesth. 2014 May;112(5):951-3. doi: 10.1093/bja/aeu127. No abstract available. PMID 24771798
- [Background] Biro P, Sermeus L, Jankovic R, Savic N, Onutu AH, Ionescu D, Godoroja D, Gurman G. Basic Features and Clinical Applicability of 'Preliminary Universal Surgical Invasiveness Score' (pUSIS): A Multi-Centre Pilot Study. Turk J Anaesthesiol Reanim. 2017 Feb;45(1):9-15. doi: 10.5152/TJAR.2017.77785. Epub 2017 Feb 1. PMID 28377835